CLINICAL TRIAL: NCT04903067
Title: An Investigation Into the Relationship Between Dietary Intake and Health-related Quality of Life in Children and Young People With Juvenile Idiopathic Arthritis
Acronym: JIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oxford Brookes University (Other)
Responsible Party: Principal Investigator, Najmeh Zare, DPhill candidate, Oxford Brookes University
Other Study IDs: 110611
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Juvenile idiopathic arthritis; children; young people; health-related quality of life; diet; physical activity
MeSH Terms: conditions — Arthritis, Juvenile; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
"Physical activity and diet in children and young people with arthritis" A qualitative study of exploring stake holder's experiences.

Juvenile Idiopathic Arthritis (JIA) is the most common type of arthritis in children under the age of 16. The disease and its therapeutic management can cause serious long-term complications, which affect general activities and quality of life. The lack of specific guidelines for safe physical activity and appropriate management of any nutritional deficit aiming our study to find out your views and opinions about the needs of children and young people with juvenile idiopathic arthritis. We want to improve our knowledge about the impact of physical activity and eating habit on juvenile idiopathic arthritis and we want to develop a tool to help evaluate care. Few studies targeting quality of life and wellbeing in children adolescent populations have adopted the diet and physical activity perspective or approaches, consequently, this research project will help to address this gap through:

1. Interview: to look at young people's current experiences with JIA as well as their parents/caregivers and health care professionals. Study findings will provide a snapshot of the current experiences of participants, helping to improve our knowledge about JIA, physical activity, and diet. Qualitative studies exploring people perspectives on their experiences, when collected systematically, adds valuable depth, insight and understanding into the issues related to JIA not possible through quantitative methodologies. This study uses a qualitative approach known as framework methodology to understand stakeholder's experience of what helps and what hinders improving the quality of life in children and young adult with JIA. 21-30 stakeholders will be recruited in Oxford UK, to take part in individual semi-structured guided interviews lasting approximately one hour. Participant responses will be transcribed by the chief investigator and analysed to extract themes that will answer the research question.
2. Delphi study: which aims to develop a diet and physical activity intervention for children and young adult with JIA.

DETAILED DESCRIPTION:
"Physical activity and diet in children and young people with arthritis" A qualitative study of exploring stake holder's experiences.

Juvenile Idiopathic Arthritis (JIA) is the most common type of arthritis in children under the age of 16. The disease and its therapeutic management can cause serious long-term complications, which affect general activities and quality of life. The lack of specific guidelines for safe physical activity and appropriate management of any nutritional deficit aiming our study to find out your views and opinions about the needs of children and young people with juvenile idiopathic arthritis. We want to improve our knowledge about the impact of physical activity and eating habit on juvenile idiopathic arthritis and we want to develop a tool to help evaluate care. Few studies targeting quality of life and wellbeing in children adolescent populations have adopted diet and physical activity perspective or approaches, consequently this research project will help to address this gap through:

1. Systematic review: to evaluate current evidence about diet, health and health related quality of life in children and young adult with JIA.
2. Interview: to look at young people's current experiences with JIA as well as their parents/caregivers and health care professionals. Study findings will provide a snapshot of current experiences of participants, helping to improve our knowledge about JIA, physical activity, and diet. Qualitative studies exploring people perspectives on their experiences, when collected systematically, adds valuable depth, insight and understanding into the issues related to JIA not possible through quantitative methodologies. This study uses a qualitative approach known as framework methodology to understand stakeholder's experience of what helps and what hinders improving the quality of life in children and young adult with JIA. 21-30 stakeholders will be recruited in Oxford UK, to take part in individual semi-structured guided interviews lasting approximately one hour. Participant responses will be transcribed by the chief investigator (PhD student) and analysed to extract themes that will answer the research question.
3. Delphi study: which aims to develop diet and physical activity intervention for children and young adult with JIA.

This protocol covers the second and third approaches only (interview and Delphi).

ELIGIBILITY:
Inclusion Criteria:

* A) Patients

  * Male or female, age range 9 to 18 years old.
  * Diagnosed with JIA.
  * Speaking and understanding English.
  * Willing and able to provide consent if 16-18 years old, or have a parent/carer to provide consent and able to provide assent if the participant is <16.
  * Having the access to telephone/video call for those who wish to have distance interview.

B) Parent/Carer

* parent or caregiver of a child with JIA.
* Willing and able to give informed consent for their own and their child's participation (if the child is under 16 years of age).
* Having the access to telephone/video call for those who wish to have distance interview.
* Speaking and understanding English. C) Healthcare professionals
* Willing and able to give informed consent.
* Clinical HCP with at least 2-year experience in treating children and young people with JIA.
* Academic in the field of clinical research in the treatment of JIA.
* Having the access to telephone/video call for those who wish to have distance interview.
* Speaking and understanding English.

Exclusion Criteria:

Individuals will be excluded from the study if ANY of the following apply:

A) Patient

* They have been diagnosed JIA but older than 18 years old.
* Unable to speak and understand English. B) Healthcare professionals
* HCP with insufficient experience in JIA management.

  * They have less than two years of managing/treating JIA patients.
  * They have worked in this field but have stopped for two years or more.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Nuffield Orthopaedic Centre Oxford, Usual referral clinic.
Sampling Method: Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
study one interviews | one hour
  views and opinions of participants

SECONDARY OUTCOMES:
study two Delphi | one hour
  consensus of views and opinions

CONTACTS AND LOCATIONS:
Locations (1):
- Najmeh Zare, Oxford, Oxfordshire, United Kingdom